CLINICAL TRIAL: NCT00978796
Title: Pilot Study Assessing Glucose Effects of Sitagliptin (Januvia) in Adult Patients With Type 1 Diabetes
Brief Title: Assessing Glucose Effects of Sitagliptin (Januvia) in Adult Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Satish K. Garg, Barbara Davis Center for Childhood Diabetes
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Merck IISP-32888; NCT01227460 (obsolete NCT alias)
Record Dates: First submitted 2009-09-14; First posted 2009-09-17 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Mellitus; Type 1 diabetes; glucose variability
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Sitagliptin Phosphate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Active Comparator): Patients will receive sitagliptin for 4 weeks and then cross over to sugar pill
  Interventions: Drug: Sitagliptin
- Sugar pill (Placebo Comparator): Subjects will receive sugar pill for 4 weeks and then cross over to active sitagliptin
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100mg tablet taken orally once daily for 4 weeks and then switch over to sugar pill taken daily for 4 weeks
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Sugar Pill — Sugar pill taken daily for 4 weeks and then switched over to active comparator of sitagliptin 100mg tablet taken daily for 4 weeks
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine the effects of sitagliptin on glucose variability both after meals and overnight in adult patients with type 1 diabetes.

DETAILED DESCRIPTION:
Improved post prandial glucose control with multiple daily injections of insulin in the DCCT study demonstrated significant reductions in microvascular complication. Similar to type 2 diabetes, patients with type 1 diabetes have a paradoxical increase in glucagon after meals which contribute to worsening post prandial glucose control. This proposed study is designed to determine if altering the glucagon axis by giving sitagliptin can improve glucose control in patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult, aged 18 to 70 years
* Type 1 diabetes mellitus as established by medical history
* Current treatment with MDI or CSII therapy for at least 3 months prior to screening visit; and using the same insulin during the last 1 month
* HbA1c ≥ 8.5%
* Subjects should routinely practice at least 2-4 blood glucose measurements per day
* BMI ≤ 35 kg/m2
* Subject must be able and willing to perform self-blood glucose monitoring and accept wearing a continuous glucose monitor for the total duration of the study
* Willing to complete a routine medical visits every 3 months
* Willing to complete a total of 7 phone visits
* Able to speak, read, and write English

Exclusion Criteria:

* On oral, inhaled or pre-mixed insulin
* On Symlin
* BMI > 35 kg/m2
* Pregnant or intends to become pregnant during the course of the study
* Severe unexplained hypoglycemia that required emergency treatment over the past 3 months
* History of hemoglobinopathies
* Diagnosis of anemia
* HbA1C greater than 12%
* Post-renal transplantation, currently undergoing dialysis, creatinine of >1.5mg/dl or a calculated creatinine clearance of <50 mL/min.
* Have extensive skin changes/diseases that inhibit wearing the sensor on normal skin
* Subjects who have a medical known allergy to adhesives
* Subjects who have an allergy to medication being used
* Currently participation in another investigational study protocol. Must have completed a previous study at least 30 days prior to being enrolled in this one
* Have any condition that, in the opinion of the Investigator, would interfere with their participation in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this pilot study is to compare 24-hour blood glucose values (overnight and pre- and post- prandial glucoses) in adult subjects with type 1 diabetes receiving either sitagliptin or placebo | Assessment done at week 4 and week 8

SECONDARY OUTCOMES:
Determine differences in fructosamine values | baseline, 4 and 8 weeks
Time spent in hypoglycemic and hyperglycemic excursions recorded on the DexCom STS continuous glucose monitor (CGM) at 3 time periods throughout the study | Assessed at week 4 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Satish Garg, MD, Principal Investigator — University of Colorado, Denver; Samuel L Ellis, Pharm.D., Principal Investigator — University of Colorado School of Pharmacy
Locations (1):
- Barbara Davis Center for Childhood Diabetes, Aurora, Colorado, United States

REFERENCES:
- [Derived] Garg SK, Moser EG, Bode BW, Klaff LJ, Hiatt WR, Beatson C, Snell-Bergeon JK. Effect of sitagliptin on post-prandial glucagon and GLP-1 levels in patients with type 1 diabetes: investigator-initiated, double-blind, randomized, placebo-controlled trial. Endocr Pract. 2013 Jan-Feb;19(1):19-28. doi: 10.4158/EP12100.OR. PMID 23186950
- [Derived] Ellis SL, Moser EG, Snell-Bergeon JK, Rodionova AS, Hazenfield RM, Garg SK. Effect of sitagliptin on glucose control in adult patients with Type 1 diabetes: a pilot, double-blind, randomized, crossover trial. Diabet Med. 2011 Oct;28(10):1176-81. doi: 10.1111/j.1464-5491.2011.03331.x. PMID 21923696